CLINICAL TRIAL: NCT04565587
Title: Rheological Characterization of the Thickener Tsururinko Quickly and Dose-response Effect on Older Patients
Brief Title: Dose-response Effect of the Thickener Tsururinko Quickly
Acronym: 58/19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morinaga Milk Industry Co., LTD (Industry)
Collaborators: Hospital de Mataró (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQUICKLY
Record Dates: First submitted 2020-08-25; First posted 2020-09-25 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Dysphagia; Dysphagia, Oral Phase; Dysphagia, Oropharyngeal; Dysphagia, Esophageal; Swallowing Disorder
Keywords: thickener; rheology; dysphagia; dose-response effect; salivary amylase effect; shear rate
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: All the participants will be assigned to the same intervention.
Masking Description: Analyisis of the therapeutic effect of the viscosities will be performed in a codified manner by a researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Videofluoroscopy (Other): All participants will undergo a Videofluoroscopy when swallowing different viscosity levels of the thickener Tsururinko Quickly (japanese thickener)
  Interventions: Other: Xanthan-gum based thickener

INTERVENTIONS:
Other: Xanthan-gum based thickener — Participants will undergo a screening procedure (V-VST) with two of the viscosities levels determined and prepared with mineral water and Tsururinko Quickly (200 and 800mPa·s). After the V-VST, a Videofluoroscopy (VFS) will be performed with thin liquid and 5 viscosity levels prepared with X-Ray contrast (Omnipaque), mineral water and Tsururinko Quickly (100, 200, 400, 800, 1600mPa·s). Participants swallow will be studied with VFS in a lateral projection and images will include the oral cavity, pharynx, larynx and cervical oesophagus. Swallows will be analysed by equipment developed to capture and digitize the swallowing sequences to assess VFS signs of safety and efficacy according to accepted definitions and to measure the timing and spatial events of the swallow response.
  Other Names: Alimentary thickener

SUMMARY:
Thickening fluids are a valid therapeutic strategy to improve safe swallowing in OD. The aim of this study is to assess the percentage of safe swallowing at different viscosity levels thickened with Tsururinko Quickly.

This study is designed to assess the therapeutic effect on safety and efficacy of swallow of Tsururinko Quickly for the levels of viscosity 100, 200, 400, 800, 1600mPa·s against thin liquid and between all the viscosity levels in older patients with Oropharyngeal Dysphagia (OD) by performing a Videofluoroscopy when swallowing. As all patients will start with thin liquid, each patient will be its own control. To analyze the effect of the salivary amylase on the thickener, participants will be asked to maintain two boluses (200 and 800mPa·s) prepared jut with mineral water in the oral cavity for 30seconds. After that period, boluses will be analyzed by a viscometer and compared to those without oral incubation.

DETAILED DESCRIPTION:
Older patients, who fulfil the eligibility criteria, are invited to participate in the study. After having signed informed consent, participants who meet the inclusion and exclusion criteria will a screening procedure (V-VST). Viscosities for the V-VST: <50, 200mPa·s and 800mPa·s. Two questions will be performed to the patient on palatability and acceptability. Palatability will be assessed by the 5-points hedonic scale and acceptability with the Scorecard - Food Action Rating Test. After it, a Videofluoroscopy (VFS) will be performed. For the VFS, participants will swallow 10mL boluses (by duplicate) of thin liquid and 5 different thickened viscosities of Tsururinko Quickly (1600, 800, 400, 200 and 100 mPa·s) with a stablished safety rule: when the subject aspirates at the first bolus of thin liquid, the second volume will not be given and the measurements will continue with the thickened varieties to the thinnest viscosity. In case the subject aspirates at one thickened bolus, the VFS ends for this specific patient. As all patients will start with thin liquid, each patient will be its own control with the non-thickened viscosity vs the others in order to establish the safety of swallow for all the levels performed. Patient's swallow will be studied with VFS in a lateral projection and images will include the oral cavity, pharynx, larynx and cervical oesophagus. After each bolus, the patient will be asked to give their opinion on the palatability of this specific bolus.

Before VFS, a bolus of 200 and 800mPa·s (without contrast) will be given to the participant in order to perform the oral incubation analysis. Participants should keep the bolus in their mouth for 30" and then spit it out. The bolus is then analysed with the viscometer at the shear rate of 50s-1 (estimated value at the oral cavity) and 300s-1 (estimated value at the pharynx). Viscosity values will be compared to the viscosity values without oral incubation. The day after the completion of the VFS participants will be asked by phone for AE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Oropharyngeal Dysphagia: clinical signs or symptoms of swallowing dysfunction (safety or efficacy impairments), based on videofluoroscopy (VFS)
* Written informed consent

Exclusion Criteria:

* No clinical signs or symptoms of swallowing dysfunction, based on videofluoroscopy (VFS)
* OD due to structural alterations
* Severe cognitive disorders or Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements and instructions
* Not able to undergo VFS due to incapability of sitting posture
* Pregnancy and/or lactating
* Allergy to any ingredient of test product or iodine products

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect on safety and efficacy of swallow of Tsururinko Quickly for the levels of viscosity 100, 200, 400, 800, 1600mPa·s against thin liquid and within each viscosity in older patients with Oropharyngeal Dysphagia (OD) | 2 days
  Percentage of participants that swallow safely (PAS score 1, 2) for each viscosity level (Rosenbek, 1996)

SECONDARY OUTCOMES:
Safety of swallowing for the levels of viscosity 100, 200, 400, 800, 1600mPa·s against thin liquid and within each viscosity in older patients with Oropharyngeal Dysphagia (OD) | 2 days
  Safety of swallowing measured by mean PAS score, percentage of patients with safe swallowing (PAS1, 2), percentage of patients with penetration (PAS score 3, 4, 5) and percentage of patients with aspiration (PAS score 6, 7, 8)
Efficacy of swallowing for the levels of viscosity 100, 200, 400, 800, 1600mPa·s against thin liquid and within each viscosity in older patients with Oropharyngeal Dysphagia (OD) | 2 days
  Efficacy of swallowing expressed by prevalence and severity of patients with oral and pharyngeal residue assessed by the scale defined by Robbins et al. 2007
Assess the effect of oral incubation with salivary amylase on Tsururinko Quickly | 2 days
  To assess the resistance of the product to the α-salivary amylase by the viscosity decrease (%)
Physiology of swallowing for the levels of viscosity 100, 200, 400, 800, 1600mPa·s against thin liquid and within each viscosity in older patients with Oropharyngeal Dysphagia (OD) | 2 days
  Swallowing physiology assessed as time to laryngeal vestibule closure (LVC) (ms), time to laryngeal vestibule opening (ms), total duration of swallowing response (ms), time to upper oesophageal sphincter opening (UESO) (ms) and bolus velocity (m/s),
Kinematics of the bolus while swallowing for the levels of viscosity 100, 200, 400, 800, 1600mPa·s against thin liquid and within each viscosity in older patients with Oropharyngeal Dysphagia (OD) | 2 days
  Kinematics of the bolus assessed as translational kinetic energy (KE; MJ) prior to entering the UES.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró, Mataró, Spain

IPD SHARING:
Plan to Share IPD: No